CLINICAL TRIAL: NCT01141647
Title: Predictive Outcome Model Over Time for Employment (PROMOTE)
Brief Title: SCI-VIP: Predictive Outcome Model Over Time for Employment (PrOMOTE)
Acronym: PrOMOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O7814-R
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Spinal Cord Injuries
Keywords: Adult; Depression; Supported Employment; Health Service; Humans; Outcomes; Quality of Life; Veterans/rh (rehabilitation); Workplace; Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries; Depression | interventions — Rehabilitation, Vocational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 24-Month Supported Employment (Experimental): Evidence-Based Supported Employment Vocational Rehabilitation or Other Vocational Services
  Interventions: Behavioral: Vocational Rehabilitation

INTERVENTIONS:
Behavioral: Vocational Rehabilitation — SCI-VIP: PrOMOTE evidence-based supported employment implemented for Veterans with spinal cord injury or other available vocational services

SUMMARY:
This study will be an extension of the Spinal Cord Injury Vocational Integration Program (SCI-VIP). The study involves research about how to help Veterans with spinal cord injury (SCI) gain employment. Vocational rehabilitation is a special field of service aimed at putting persons with disabilities in the best possible position to become employed. The Veterans Administration has a long history of providing vocational rehabilitation for Veterans with mental health issues and has recently started providing similar services to persons with physical disabilities, including SCI. Past research has shown that vocational rehabilitation is effective in helping some Veterans with spinal cord injury (SCI) gain employment. The extension of this work through PrOMOTE study will establish a large national database of over 2000 Veterans with SCI, containing extensive employment, medical, functional and psychosocial data. The study will analyze both quantitative and qualitative measures to maximize its findings.

DETAILED DESCRIPTION:
Extending SCI-VIP through PrOMOTE will operationalize the critical features of supported employment that lead to obtaining and maintaining employment over time in spinal cord injury. There are no current studies that examine how the level and intensity of supported employment services by Veterans with SCI impacts employment outcomes. This extension will allow the examination of longitudinal factors associated with successful employment that are not possible within the time constrains of SCI-VIP and to extend the cost-effectiveness analysis and budget impact analysis to include longer term and costs of quality of life outcomes. The study will include a more comprehensive qualitative analysis across several sites of factors that contribute to program success. The PrOMOTE study will add three more sites. This expansion will allow examination of outcomes in areas where there is a high penetration of OIF/OEF Veterans as well as sites where there are other vocational programs available.

Primary HO: Identify factors that predict employment after SCI.

Secondary HO 1: Determine ongoing effectiveness of SE over time.

Secondary HO 2: Evaluate the effectiveness of implementation strategy and level of SE model implementation across sites.

Secondary HO 3: Determine costs, health care utilization over time and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

All Veterans who meet inclusion criteria will be approached about completing a baseline interview to gather information on employment, health, and quality of life after spinal cord injury.

Inclusion criteria for the baseline interview include:

* 18 to 65 years old
* Spinal Cord Injury
* Medically and neurologically stable

At the end of the baseline interview, some of these Veterans who meet additional inclusion criteria will be enrolled to receive the SE intervention or other available vocational services and complete longitudinal follow-up interviews every three months while participating in the study.

The additional inclusion criteria for enrollment in vocational services include:

* Unemployed
* Living within 100 mile radius of the enrolling VA Medical Center
* Desiring competitive employment

A subsample of Veterans who consent to the study will be selected for participation in qualitative interviews. Family members and/or caregivers identified by these Veterans may also be included in qualitative interviews. A representative sample of VA staff members who provide care to these Veterans will also be approached to participate in qualitative interviews.

Exclusion Criteria:

* Medically and/or surgically unstable
* Mentally impaired such that independent reasoning and judgment jeopardize safety of self or others
* Active alcohol and/or drug dependency that is untreated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1047 (Actual)
Dates: Start 2011-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ottomanelli, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (7):
- United States (7):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
Data will only be presented de-identified.

REFERENCES:
- [Result] Cotner BA, Njoh EN, Trainor JK, O'Connor DR, Barnett SD, Ottomanelli L. Facilitators and barriers to employment among veterans with spinal cord injury receiving 12 months of evidence-based supported employment services. Top Spinal Cord Inj Rehabil. 2015 Winter;21(1):20-30. doi: 10.1310/sci2101-20. PMID 25762857
- [Result] Sutton BS, Ottomanelli L, Njoh E, Barnett SD, Goetz LL. The impact of social support at home on health-related quality of life among veterans with spinal cord injury participating in a supported employment program. Qual Life Res. 2015 Jul;24(7):1741-7. doi: 10.1007/s11136-014-0912-4. Epub 2015 Jan 11. PMID 25577499
- [Derived] Goetz LL, Ottomanelli L, Barnett SD, Sutton B, Njoh E. Relationship Between Comorbidities and Employment Among Veterans with Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2018 Winter;24(1):44-53. doi: 10.1310/sci16-00047. Epub 2017 Sep 27. PMID 29434460
- [Derived] Budd MA, Dixon TM, Barnett SD, Njoh E, Goetz LL, Ottomanelli L. Examination of traumatic brain injury exposure among veterans with spinal cord injury. Rehabil Psychol. 2017 Aug;62(3):345-352. doi: 10.1037/rep0000129. Epub 2017 Jun 8. PMID 28594193
- [Derived] Ottomanelli L, Goetz LL, Barnett SD, Njoh E, Dixon TM, Holmes SA, LePage JP, Ota D, Sabharwal S, White KT. Individual Placement and Support in Spinal Cord Injury: A Longitudinal Observational Study of Employment Outcomes. Arch Phys Med Rehabil. 2017 Aug;98(8):1567-1575.e1. doi: 10.1016/j.apmr.2016.12.010. Epub 2017 Jan 20. PMID 28115071

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1047 subjects were enrolled; 450 were ineligible for supported employment (SE) services and 318 were out of the SE recruitment window. 279 SE participants remained, and 66 were analyzed separately because of their previous participation in SE. For the purposes of reporting 213 subjects were included
Groups:
- 24-Month Supported Employment: Evidence-based supported employment implemented for Veterans with spinal cord injury or other available vocational services
Period: Overall Study
Arm/Group | 24-Month Supported Employment
Started | 213
Completed | 167
Not Completed | 46

BASELINE CHARACTERISTICS:
Arm/Group | 24-Month Supported Employment
Number analyzed (Participants) | 1047
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1047
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 1002
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasion | 653
  African American | 306
  Asian | 13
  Native American | 15
  Other/Unknown | 60
Functional Independence Measure [Mean (Standard Deviation); unit: units on a scale] — This measure contains 18 items composed of 13 motor-related tasks and 5 cognitive-related tasks. Each task is rated on a 7-point ordinal (1=total assistance (or complete dependence) to 7=complete independence). The range of scores is 18 to 126, with the lower score indicating greater dependence.
  units on a scale | 71.5 (27.2)
ASIA Impairment Scale (AIS) [Number; unit: participants] — ASIA Impairment is used to describe an individual's functional level impairment due to spinal cord injury. Ranging from level A indicating greatest impairment to level E all functioning having returned.
  participants
    A | 408
    B | 121
    C | 133
    D | 366
    E | 7
    Missing | 12
AIS and neurological Level [Number; unit: participants] — High Tetraplegia, AIS, A, B, C: high cervical injury with upper and lower extremities motor and/or sensory impairment.
  Low Tetraplegia, AIS, A, B, C low cervical injury with upper and lower extremities motor and/or sensory impairment.
  Paraplegia, AIS, A, B,C: an injury to the thoracic or lumbar area of the spinal cord resulting in motor and/or sensory impairment of the lower extremities.
  Tetraplegia or Paraplegia AIS D/E: cervical, thoracic or lumbar injury with the least amount of motor and/or sensory impairment.
  participants
    High Tetraplegia, AIS, A, B, C | 91
    Low Tetraplegia, AIS A,B,C | 200
    Paraplegia, AIS A,B,C | 371
    AIS D/E | 372
    Missing | 13
Marital Status [Number; unit: participants]
  Married | 373
  Divorced | 366
  Other | 305
  Refused/NA | 3
Education Years [Mean (Standard Deviation); unit: years] | 13.8 (2.4)
VA Benefits Recipient [Number; unit: participants]
  Yes | 655
  No | 369
  N/A | 2
  Missing/Other | 21
Military Service-connected benefits for SCI [Number; unit: participants] — Service connected disability compensation is a monetary benefit paid to Veterans who are determined by VA to be disabled by an injury or illness that was incurred or aggravated during active military service. The level of benefit is indicated as a percentages in intervals of 10 starting at 0. Ratings of 10% or higher are monetarily compensated. To be Spinal Cord Injury service connected 100% is the highest level of compensation for a SCI that was incurred or aggravated during active military service.
  participants
    Yes | 331
    No | 237
    N/A | 444
    Missing/Other | 35
Military Service-connected 100% [Number; unit: participants]
  Yes | 341
  No | 258
  N/A | 379
  Missing | 69
Non-Service-connected pension [Number; unit: participants]
  Yes | 132
  No | 498
  N/A | 378
  Missing/Other | 39
Monthly Non-Service-connected pension [Mean (Standard Deviation); unit: Dollars] | 1078 (795.4)
Monthly Social Security Income Benefits [Mean (Standard Deviation); unit: Dollars] | 994 (485.2)
Monthly Social Security Disability Insurance Benefits [Mean (Standard Deviation); unit: Dollar] | 1215 (556.2)
Neither Social Security Income/Social Security Disability Insurance Recipient [Number; unit: participants]
  Neither | 234
  One or more | 798
  N/A | 2
  Missing/Other | 13
Measures of Handicap (CHART) [Mean (Standard Deviation); unit: units on a scale] — The CHART is a tool assessing an individuals level of handicap with six subscales. It consists of 32 items which assess six dimensions (cognitive independence, physical independence, mobility, occupation, social integration, and economic self-sufficiency). The scores for each subscale range from 0-100, with a score of 100 indicates no handicap in a given dimension.
  units on a scale
    Social Integration | 88.6 (14.5)
    Occupation | 47.6 (33.9)
    Mobility | 76.8 (23.9)
    Physical | 85.4 (20.9)
    Cognitive | 90.7 (16.2)
    Economic Self Sufficiency | 57.9 (42.1)
Quality of Life VR-36 [Mean (Standard Deviation); unit: T-score] — The VR-36 is used to measure health related quality of life. Assesses 8 domains (general health, physical functioning, role limitations, pain, energy-fatigue, social functioning and mental health). The 36 items have a 5-point ordinal response and result in providing two scores, physical component score (PCS) and mental component score (MCS). Items are summed with a range of 0-100. The PCS and MCS are standardized using a T-score and normed to a U.S. population (1990 population) score of 50 and standard deviation of 10.Higher scores means better outcome.
  T-score
    Mental Component Scale | 56.5 (12.4)
    Physical Component Scale | 27.2 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Identify Factors That Predict Employment After SCI.
Description: To model the probability of obtaining CE, we first dichotomized CE as 'yes' or 'no'. The Competitive Employment Rate is reported in Outcome Measure 2. We then used unconditional logistic regression to model the probability of obtaining CE through a univariate modeling approach to determine statistically significant predictors of CE. Statistically significant predictors at the p<0.10 criterion level were then explored in a final multivariate model. Demographic (age, race, marital status, etc.), clinical (severity of injury, comorbidities, time since injury, etc.), barriers and facilitators, and quality of life (depression, Satisfaction with Life, etc.) were considered for modeling. A final model was obtained by including all parameters meeting the p<0.10 criterion into a final multivariate model.
Time Frame: 24-month phase with face-to-face quarterly interviews
Measure: Number (90% Confidence Interval); unit: Odds Ratio
Groups:
- 24-Month Supported Employment: Participants in Supported Employment.
Arm/Group | 24-Month Supported Employment
Number analyzed (Participants) | 213
Odds Ratio | 3.56 [1.80 to 7.07]
Statistical Analysis 1: Comparison: 24-Month Supported Employment; Test type: Superiority or Other; Odds Ratio (OR) = 3.56, 90% CI 2-sided [1.80 to 7.07]

2. Secondary Outcome: Employment Rate
Description: Competitive Employment (CE) rate for individuals who participated in the Supported Employment arm of the PrOMOTE Study.
Time Frame: 24 Months
Measure: Number; unit: percentage of participants with CE
Arm/Group | 24-Month Supported Employment
Number analyzed (Participants) | 213
percentage of participants with CE | 43.2

3. Secondary Outcome: Determine Ongoing Effectiveness of SE Over Time.
Description: This measure is used to evaluate the participants who were both in SCI-VIP and PrOMOTE. It assesses the number of people who obtained CE in SCI-VIP and sustained the same CE through their time in the PrOMOTE study. The cohort of SCI-VIP SE participants in PrOMOTE were analyzed separately from the 213 PrOMOTE participants.
Time Frame: 48-month phase with face-to-face quarterly interviews
Population: Number of participants in 24-month SE and 24-month SCI-VIP (previous study).
Measure: Number; unit: participants
Groups:
- 48-Month Supported Employment: Evidence-Based Supported Employment Vocational Rehabilitation or Other Vocational Services
  Vocational Rehabilitation: SCI-VIP: PrOMOTE evidence-based supported employment implemented for Veterans with spinal cord injury or other available vocational services
Arm/Group | 48-Month Supported Employment
Number analyzed (Participants) | 30
participants | 5

4. Secondary Outcome: Evaluate the Effectiveness of Implementation Strategy and Level of SE Model Implementation Across Sites.
Description: Level of implementation was assessed by interviewing clinical and vocational providers from the seven sites who were involved in or knowledgeable about the program. Values reported represent the numbers of clinical staff who cited having the VRS integrated on the clinical team, a full-time VRS, leadership support, engagement of staff, resources provided immediately, making adjustments to the implementation to fit with the local context, and having audit and feedback as supporting strong implementation
Time Frame: 24-month phase with face-to-face quarterly interviews
Population: Each stage comprised of two site visits. Please note that in the early stage fit of IPS model and audit and feedback were not assessed in either of the site visits, hence a value of zero is entered. Also note that in the late stage obtaining resources, fit of IPS model, and audit and feedback were only assessed at 1/2 of the site visits.
Measure: Number; unit: participants
Groups:
- Early Stage: Interview data from clinical staff during year 1.
- Mid Stage: Interview data from clinical staff from year 2.
- Late Stage: Interview data from clinical staff in year 3.
Arm/Group | Early Stage | Mid Stage | Late Stage
Number analyzed (Participants) | 43 | 40 | 36
participants
  Integration of vocational and clinical team | 32 | 30 | 30
  VRS | 20 | 14 | 19
  Leadership Support | 17 | 17 | 13
  Engagement of staff | 21 | 9 | 13
  Obtaining resources | 10 | 9 | 6
  Fit of IPS Model | 0 | 13 | 4
  Audit and Feedback | 0 | 0 | 7

5. Secondary Outcome: Determine Total Cost Per Patient Over 24 Months
Description: Total cost is the mean total cost per patient over 24 months in US dollars. The minimum value is 0 representing no cost in US dollars and larger numbers indicating higher costs in US dollars.
Time Frame: 24-month phase with face-to-face quarterly interviews
Population: 213 SE participants in the PrOMOTE study were compared to 76 individuals in the control group of the SCI-VIP study.
Measure: Mean (Standard Deviation); unit: US dollars
Groups:
- Participants in SCI-VIP Standard Care: Standard Care group from SCI-VIP trial (NCT00117806): Standard care varies slightly between participating VA SCI centers, however, usually involves referral outside SCI center
Arm/Group | 24-Month Supported Employment | Participants in SCI-VIP Standard Care
Number analyzed (Participants) | 213 | 76
US dollars | 134,029 (148,449) | 169,433 (187,661)

6. Secondary Outcome: Determine Cost-effectiveness.
Description: QALYs are the mean quality adjusted life years per patient for the Supported Employment and Standard Care groups. The QALY is a non-negative number assessing the quality and length of life and not just the crude number of years. The minimum value is 0 representing no improvement in the quality of life or length of life and larger numbers indicate healthier and longer life. Maximum QALYs are limited only by the life span of study participants, but may not exceed 1 (perfect health) in any given year.
Time Frame: 24-month phase with face-to-face quarterly interviews
Population: 213 SE participants in the PrOMOTE study were compared to 76 individuals in the control group of the SCI-VIP study.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | 24-Month Supported Employment | Participants in SCI-VIP Standard Care
Number analyzed (Participants) | 213 | 76
years | 1.27 (0.068) | 1.15 (0.058)

ADVERSE EVENTS:
Time Frame: 4 years
Description: Reports provided to the coordinating center by site coordinators at each of the project's seven sites. All reported events were determined by the local IRBs to be unrelated to the study.
Groups:
- Baseline Sample (N=1047): Evidence-Based Supported Employment Vocational Rehabilitation or Other Vocational Services
  Vocational Rehabilitation: SCI-VIP: PrOMOTE evidence-based supported employment implemented for Veterans with spinal cord injury or other available vocational services
Arm/Group | Baseline Sample (N=1047)
Serious Adverse Events (participants affected / at risk) | 150/1047
Other Adverse Events (participants affected / at risk) | 21/1047
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Sample (N=1047) (N=1047)
Hospitalization (Blood and lymphatic system disorders) | 1 (1)
Hospitalization (Cardiac disorders) | 2 (2)
Hospitalization (Gastrointestinal disorders) | 5 (5)
Hospitalization (Immune system disorders) | 2 (2)
Hospitalization (Infections and infestations) | 33 (45)
Hospitalization (Injury, poisoning and procedural complications) | 14 (16)
Hospitalization (Investigations) | 5 (7)
Hospitalization (Metabolism and nutrition disorders) | 2 (3)
Hospitalization (Musculoskeletal and connective tissue disorders) | 1 (2)
Hospitalization (Nervous system disorders) | 7 (7)
Hospitalization (Psychiatric disorders) | 8 (10)
Hospitalization (Renal and urinary disorders) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hospitalization (Skin and subcutaneous tissue disorders) | 9 (12)
Hospitalization (Social circumstances) | 7 (9)
Hospitalization (Surgical and medical procedures) | 38 (50)
Hospitalization (Vascular disorders) | 1 (1)
Life Threatening (Psychiatric disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Other important medical event (Infections and infestations) | 1 (1)
Other important medical event (Musculoskeletal and connective tissue disorders) | 1 (1)
Incarceration (Social circumstances) | 1 (1)
Death (Cardiac disorders) | 3 (3)
Death (Infections and infestations) | 6 (6)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Death (Nervous system disorders) | 27 (27)
Death (Psychiatric disorders) | 1 (1)
Death (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Death (Skin and subcutaneous tissue disorders) | 1 (1)
Death (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Sample (N=1047) (N=1047)
Hospitalization - Respite (Social circumstances) | 14 (21)
Hospitalization - Annual Exam (Surgical and medical procedures) | 7 (8)

LIMITATIONS AND CAVEATS:
Majority of sample is male.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes